CLINICAL TRIAL: NCT07050862
Title: Circuity-guided Repetitive Transcranial Magnetic Stimulation (rTMS) for Tobacco Use in Veterans: A Comparison of Insula-rTMS and Prefrontal-rTMS
Brief Title: rTMS for Tobacco Use in Veterans
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NURA-005-24F; Pro00141919 (Other: IRB Approval ID)
Record Dates: First submitted 2025-05-15; First posted 2025-07-03 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Tabacco Use Disorder; rTMS
Keywords: Tabacco; substance abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Standard rTMS vs Precision rTMS
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Deep rTMS (Active Comparator): DThe first group will receive 10 Hz DTMS (standard TMS) with a protocol of 3 seconds on, 15 seconds off, and a total of 1800 pulses/session, lasting 18 minutes, targeting the bilateral insula and lateral prefrontal cortex.
  Interventions: Device: Transcranial Magnetic Stimulation
- Precision TMS (Experimental): The other group will receive 10 Hz personalized-image-guided and Efield-modeling dose rTMS (precision TMS) with a protocol of 5 seconds on, 10 seconds off, and a total of 3000 pulses/session, lasting 15 minutes, targeting the left DLPFC.
  Interventions: Device: personalized-image-guided and E-field-modeling dose rTMS (precision TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The first group will receive 10 Hz DTMS (standard TMS) with a protocol of 3 seconds on, 15 seconds off, and a total of 1800 pulses/session, lasting 18 minutes, targeting the bilateral insula and lateral prefrontal cortex.
  Other Names: Deep TMS, Standard rTMS
  Arms: Deep rTMS
Device: personalized-image-guided and E-field-modeling dose rTMS (precision TMS) — with a protocol of 5 seconds on, 10 seconds off, and a total of 3000 pulses/session, lasting 15 minutes, targeting the left DLPFC.
  Arms: Precision TMS

SUMMARY:
Cigarette smoking is a significant public health concern for Veterans. Encouraging smoking cessation continues to be a top priority for the Veterans' Administration as Veterans who use tobacco experience negative health effects, including cancer, heart disease, and mental disorders. Despite the efficacy of current evidence-based pharmacotherapies and psychotherapies for smoking cessation, alternative treatments are critically needed. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive form of brain stimulation, US FDA-approved for smoking cessation. In this protocol, the investigators propose comparing the two rTMS protocols (standard TMS vs. precision TMS) to find a better treatment parameter for smoking cessation in Veterans. Identifying an efficacious rTMS protocol would benefit Veterans who want to quit smoking.

DETAILED DESCRIPTION:
Cigarette smoking rates are high, and quitting rates are lower in the Veteran population in the United States compared to the nonveteran population. In addition, Veterans report being more likely to have smoking- related illnesses and morbidity. Despite the efficacy of current evidence-based pharmacotherapies and psychotherapies for smoking cessation, alternative treatments are critically needed. Repetitive transcranial magnetic stimulation (rTMS), has already displayed remarkable potential for producing novel, non- pharmacological interventions for neuropsychiatric disorders, including tobacco use disorder (TUD). The group's studies demonstrate that 10 Hz rTMS over the left dorsolateral prefrontal cortex (DLPFC) reduced cue craving and cigarette consumption and increased quit rate. Instead of stimulating the superficial cortex, deep TMS (DTMS) has been permitted to target deep brain structures such as the insula. DTMS has also been approved to reduce cigarette consumption and increase quit rate and was FDA-approved as a treatment option for TUD. Neuroimaging techniques such as functional magnetic resonance imaging (fMRI) have provided insight into the neurocircuitry of TUD and its therapeutic effect for smoking cessation. Recently, the investigators' team completed an image-guided randomized controlled trial (RCT) study to compare 10 Hz rTMS over the left DLPFC to 1 Hz over the medial orbitofrontal cortex (mOFC) and sham in healthy smokers. The results showed that 10 Hz over DLPFC rTMS reduced cigarette consumption more than 1 Hz mOFC and sham. In addition, 10 Hz DLPFC rTMS increased brain activity in DLPFC and decreased brain activity in mOFC. The findings suggested that the effect of rTMS depended on the different brain regions of stimulation. To date, the efficacy of rTMS for smoking cessation has not yet been evaluated in Veterans. In this protocol, the investigators propose comparing the two rTMS protocols (DTMS vs. image-guided TMS) to find a better treatment parameter for smoking cessation in Veterans. Targeting two candidate brain regions (DLPFC vs. insula) with two different TMS treatment parameters will be performed. This application aims to identify a better rTMS treatment for smoking cessation and further develop a circuit-based precision rTMS therapy for TUDs in Veterans. The investigators hypothesize that image-guided DLPFC TMS (precision TMS) treatment will produce superior effects than insula DTMS (standard TMS) in reducing cigarette consumption. The investigators will also determine that image-guided DLPFC increases the connectivity between DLPFC, mOFC, and nucleus accumbens (NAc). In the 4-year study, the investigators will recruit 56 treatment-seeking TUDs. Participants will be randomized into two groups: The first arm is 10Hz rTMS (1800 pulses/session) over the bilateral insula with FDA-cleared DTMS (H4-coil). The other arm is image-targeted 10 Hz rTMS over the left DLPFC with figure 8 coil (3000 pulses/session). Both rTMS treatments will include 15 daily rTMS treatments for 3 weeks and 3 weeks of once- weekly rTMS. The primary endpoint will be the reduction of cigarette consumption at the end of the 3-week rTMS treatment. Aim 1: Determine whether precision image-guided TMS over the left DLPFC results in a larger reduction in cigarette consumption compared to standard DTMS targeting the insula. The primary outcome will be cigarettes per day during the treatment course. The investigators will compare the reduction of cigarette compensation between two treatment groups at the end of the 3-week rTMS treatment. Aim 2: Determine whether precision image-guided TMS increases activity in the DLPFC and modulates connectivity among the DLPFC, mOFC, and NAc and whether standard DTMS increases activity in the insula, [mOFC] and modulates connectivity among the insula, [mOFC] and NAc. The investigators will compare precision TMS to standard TMS using whole-brain imaging and network connectivity analyses. Aim 3 (exploratory): Determine whether the reductions in cigarette consumption are associated with the modulated connectivity among DLPFC, [mOFC] and NAc after precision TMS and the modulated connectivity among insula, [mOFC] and NAc after standard TMS. The investigators will test if brain connectivity can be used to predict the clinical effects of rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Males and females between the ages of 18 and 70
* Individuals who smoke 10 or more cigarettes per day and have a CO level > 10 ppm indicative of recent smoking
* Those who have not received substance abuse treatment within the previous 30 days
* Those who have been stable on psychotropic medications for at least three months
* For females, those who test non-pregnant and use adequate birth control
* Those who are willing to provide informed consent
* Those who can comply with protocol requirements and likely complete all study procedures
* Those who are motivated to quit smoking (based on responses of "very likely" or "somewhat likely" in the motivation questionnaire

Exclusion Criteria:

* Current moderate to severe substance use of any psychoactive substances other than nicotine or caffeine, as defined by DSM-V criteria
* Contraindications to MRI (e.g., metal in the skull, orbital or intracranial cavity, or claustrophobia)
* Contraindications to rTMS (history of a seizure or epilepsy)
* A history of autoimmune, endocrine, viral, or vascular disorders affecting the brain
* History or MRI evidence of neurological disorder that would lead to local or diffuse brain lesions or significant physical impairment
* Unstable cardiac disease, uncontrolled hypertension, severe renal or liver insufficiency, or sleep apnea
* Major Axis I disorders diagnosed according to DSM-V criteria, such as bipolar affective disorder, schizophrenia, dementia, or major depression

  * Regarding the Veteran population, we will enroll smokers who have PTSD
* Current use of other forms of nicotine delivery, such as nicotine patches or electronic cigarettes
* Currently prescribed bupropion and/or varenicline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Cigarettes per day | The cigarettes per day will be measured up to 3 weeks for the outcome 1
  The investigators will compare the reduction of cigarette consumption between the two treatment groups at the end of the 3-week rTMS treatment. A higher reduction of CPD means a better treatment result.
Brain Imaging Outcomes - Cue Craving Scans | 3-weeks
  fMRI scans of all Veterans to look at brain function connectivity. The investigators will compare the changes of brain activity between two treatment conditions.

SECONDARY OUTCOMES:
7-day continuous quit rate (CQR) | 10 week
  Abstinence during a consecutive 7-day period in the treatment stage
Likert Visual Analog Cue Craving Scale | 10 weeks
  Assess changes in subjective craving with each session. The visual analog cue craving scale from 0 to 7. 0 = minimum, 7 = maximum. A higher score means more craving (worse).
Fagerstrom Test for Nicotine Dependence (FTND) | 10 weeks
  Standardized tool to assess intensity of physical addiction to nicotine.
Minnesota Nicotine Withdrawal Scale-Revised | 10 weeks
  Self-report scale developed to evaluate the severity of nicotine withdrawal symptoms. self-report scale developed to evaluate the severity of nicotine withdrawal symptoms. It includes 15 items. Each item is from 0 to 4, total score, 0 = minimum, 60 = maximum. A higher score means worse.
Questionnaire of Smoking Urges- Brief (QSU-B ) | 10 weeks
  A brief 10-item scale assessing smoking urges. There are 10 questions. Each question can be rated from 1 to 7. Total score: 10 is minimum, 70 is maximum. A higher score means worse.
Cabry Oxy levels | 3-week
  0-6 ppm: no smoker, 7-19 ppm: light smoker; 20 or more ppm: heavy smoker.
Biomarkers | 10 week
  Urine cotinine levels will be measured. Urine creatinine will also be measured for the correction of urine cotinine. Urine cotinine levels will be measured. Urine creatinine will also be measured for the correction of urine cotinine. A higher level is worse.
PTSD Checklist for DSM-5 | 10 week
  20 item self report measure to assess DSM-5 PTSD. It includes 20 items. Each item will rate from 0 to 4. Minimum = 0, Maximum = 80. A higher score means worse.
Patient Health Questionnaire (PHQ-9), | 10-weeks
  PHQ-9 is a self-report that screens for depression and measures its severity.
Generalized-Anxiety-Disorder (GAD- 7) | 10 week
  7 item scale that screens for and assess severity of GAD. There are 7 question in the scale. Each question can be 0 to 3. Minimum = 0, Maximum = 27. A higher scores mean worse.

CONTACTS AND LOCATIONS:
Overall Officials: Xingbao Li, MD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li X, Hartwell KJ, Henderson S, Badran BW, Brady KT, George MS. Two weeks of image-guided left dorsolateral prefrontal cortex repetitive transcranial magnetic stimulation improves smoking cessation: A double-blind, sham-controlled, randomized clinical trial. Brain Stimul. 2020 Sep-Oct;13(5):1271-1279. doi: 10.1016/j.brs.2020.06.007. Epub 2020 Jun 10. PMID 32534252
- [Background] Li X, Hartwell KJ, Owens M, Lematty T, Borckardt JJ, Hanlon CA, Brady KT, George MS. Repetitive transcranial magnetic stimulation of the dorsolateral prefrontal cortex reduces nicotine cue craving. Biol Psychiatry. 2013 Apr 15;73(8):714-20. doi: 10.1016/j.biopsych.2013.01.003. Epub 2013 Feb 26. PMID 23485014
- [Background] Li X, Toll BA, Carpenter MJ, Nietert PJ, Dancy M, George MS. Repetitive Transcranial Magnetic Stimulation for Tobacco Treatment in Cancer Patients: A Preliminary Report of a One-Week Treatment. J Smok Cessat. 2022 Jul 11;2022:2617146. doi: 10.1155/2022/2617146. eCollection 2022. PMID 35909440